CLINICAL TRIAL: NCT03430401
Title: Computer-based Cognitive Rehabilitation Program to Improve Cognition and Delay Deterioration in Functional Performance for Healthy Older Adults, Older People With Mild Cognitive Impairment and Mild Dementia
Brief Title: Computer-based Cognitive Rehabilitation Program for Healthy Older Adults, Older People With Mild Cognitive Impairment and Mild Dementia
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Western Sydney (Other)
Responsible Party: Principal Investigator, Karen Liu, Associate Professor, University of Western Sydney
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: UWesternSydney
Record Dates: First submitted 2018-02-05; First posted 2018-02-12 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Mild Cognitive Impairment; Mild Dementia; Healthy Older Adults
Keywords: memory encoding; functional performance
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Perceptual-based memory encoding (Experimental): It will involve the use of visual imagery and the method of loci. To achieve this, each of the 15 daily tasks will be filmed and a short video created. In addition, each task will be broken down into 5-6 photographed steps based on activity analysis and task breakdown. The program will prompt the user to indicate in which room of the house the task would usually be completed. Once correct location is identified, the program will prompt the user to watch a chosen daily task video and then visualise themselves completing the task in their home environment.
  Interventions: Behavioral: Perceptual-based memory encoding
- Semantic-based memory encoding (Experimental): It will incorporate association-based strategies to assist with recalling the steps of daily tasks. The steps of a given daily task will be provided and the user will be prompted to link the steps using a honeycomb concept, which makes use of the chunking method to encode the sequenced steps. Following this, the program will prompt the user to categorise the steps according to their association with given words cues. The word cues will represent time, places, objects, and people. The program will then take the user response and form a verbal and visual story according to the responses given. The program will help identify any problems in the sequencing and prompt the user to re-categorise if required.
  Interventions: Behavioral: Semantic-based memory encoding
- Cognitive stimulation (Active Comparator): Participants will complete an online cognitive exercise program, Lumosity (Sarkar, Scanlon, & Drescher, 2007). A study conducted by Hardy, Drescher, Sarkar, Kellett, and Scanlon (2011) indicated that participants who engaged in Lumosity showed greater improvements in memory in comparison to a non-intervention control group.
  Interventions: Behavioral: Cognitive stimulation

INTERVENTIONS:
Behavioral: Perceptual-based memory encoding — It will run for 12 weeks with a 1-hour training session each week, supervised by a rehabilitation professional.
  In addition, two 30-minute home-based training sessions will be completed by participants. In the home training session, participants will practice specific daily tasks that are covered in the previous professional-led session through the use of the computer-based intervention.
  Arms: Perceptual-based memory encoding
Behavioral: Semantic-based memory encoding — It will run for 12 weeks with a 1-hour training session each week, supervised by a rehabilitation professional.
  In addition, two 30-minute home-based training sessions will be completed by participants. In the home training session, participants will practice specific daily tasks that are covered in the previous professional-led session through the use of the computer-based intervention.
  Arms: Semantic-based memory encoding
Behavioral: Cognitive stimulation — The frequency, duration and the number of sessions will be consistent with the experimental interventions.
  Arms: Cognitive stimulation

SUMMARY:
This study will adopt a newly developed computer-based cognitive rehabilitation program targeting the encoding stage of memory. The aims of the study are:

1. To test the feasibility of conducting a newly developed computer-based cognitive rehabilitation program for healthy older adults, people with MCI and mild dementia.
2. To test the effectiveness of the newly developed program in improving cognitive function and enabling maintenance of occupational performance in healthy older adults, people with MCI or mild dementia.

Using an iPad application, study participants will learn a memory encoding strategy to support completion of their daily activities. By implementing memory encoding strategies during the mild stages of cognitive decline, the project aims to prolong independence in functional performance. It is anticipated that adoption of the same memory strategies will enable maintain performance as they may experience ongoing cognitive decline.

DETAILED DESCRIPTION:
This study extends on the positive results of a pilot study (Lim et al., 2012) which demonstrated the effectiveness of a cognitive training program combined with perceptual and semantic memory encoding strategies. Following the intervention phase of the pilot study, elements of cognition were examined using standardised assessments. The participants showed improved general attention (p = 0.03), memory (p = 0.03) and cognitive function including naming (p = 0.02), construction (p = 0.01), memory (p = 0.02) and similarities (p = 0.001) all of which are necessary for functioning in daily activities. However, due to the combination of strategies used during the pilot study, the isolated effect of perceptual and semantic memory encoding strategies could not be determined. It has been found that the effects of aging impact negatively on both semantic and perceptual encoding. However, with age, there tends to be a greater impact on an individual's ability to use perceptual encoding strategies in comparison to those of semantic (Kuo, Liu, Ting, & Chan, 2014). This varies in the case of individuals in the early stages of Alzheimer's disease in which many individuals will show progressive impairment in semantic memory (Hodges & Patterson, 1995). As dementia has been positively correlated with Mild Cognitive Impairment (MCI) but not often diagnosed until much later in the course of the disease and as not all individuals with MCI will progress to dementia it would be beneficial prior to undertaking a memory encoding intervention program to understand if an individual would benefit greater from undertaking a semantic or a perceptual memory encoding rehabilitation approach. Although it may be easy for a healthy adult to report their preference in encoding style, an individual with MCI or mild dementia may find this more difficult due to the abstract complexity of the concepts. As it is known that not all cases of MCI progress to dementia, this study aims at identifying if individuals with MCI or mild dementia will benefit from intervention based on both semantic and perceptual encoding styles.

In addition, given the benefit and successful use of computer-based programs in elderly, this study will develop the memory encoding training program into a user-friendly computer-based program in healthy older adults, older adults with MCI or mild dementia will be able to use under the guidance of rehabilitation professionals.

ELIGIBILITY:
Selection Criteria for healthy older adults:

1. Score greater than 24 on the Mini-Mental State Examination, 2nd edition, standard version (MMSE)
2. Score less than 5 on the 15-item Geriatric Depression Scale - Short Form (GDS)
3. No diagnosis of probable dementia (as per NINCDS-ADRDA Alzheimer's Criteria); and
4. Are able to provide voluntary consent to participate in the study.

Selection Criteria for people with MCI:

1. No diagnosis of probable dementia (as per NINCDS-ADRDA Alzheimer's Criteria);
2. Have a Clinical Dementia Rating Score (CDR) of 0 indicating no dementia;
3. Meets the diagnostic criteria for MCI (Petersen, 2004); and
4. Are able to provide voluntary consent to participate in the study.

Selection Criteria for people with mild dementia:

1. Have a diagnosis of probable dementia;
2. Have a CDR score of 1 indicating mild dementia;
3. Have a career or family members who are able to report functional performance; and
4. Are able to provide voluntary consent to participate in the study, or have a guardian to provide consent.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Disability Assessment for Dementia - Change from baseline after the intervention | Baseline and after the intervention (12 weeks)
Lawton and Brody Instrumental Activities of Daily Living Scale - Change from baseline after the intervention | Baseline and after the intervention (12 weeks)

SECONDARY OUTCOMES:
Color Trails Test - Change from baseline after the intervention | Baseline and after the intervention (12 weeks)
Repeatable Battery for the Assessment of Neuropsychological Status - Change from baseline after the intervention | Baseline and after the intervention (12 weeks)
Behavior Rating Inventory of Executive Function - Change from baseline after the intervention | Baseline and after the intervention (12 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Karen P.Y. Liu, PhD, Principal Investigator — Western Sydney University
Locations (1):
- Western Sydney University, Penrith, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tulliani N, Bye R, Bissett M, Coutts S, Liu KPY. The feasibility and acceptability of an app-based cognitive strategy training programme for older people. Pilot Feasibility Stud. 2023 Jun 30;9(1):109. doi: 10.1186/s40814-023-01334-x. PMID 37391842